CLINICAL TRIAL: NCT03098810
Title: Effect of Zinc Supplementation on Appetite and Growth of Primary Malnourished Children
Brief Title: Effect of Zinc Supplementation on Appetite and Growth in Primary Malnourished Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marian girgis, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2272009
Record Dates: First submitted 2017-03-02; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Appetite Disorders
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal children (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- Malnourished children (Experimental): Oral zinc sulphate syrup
  Interventions: Drug: Zinc sulphate

INTERVENTIONS:
Drug: Zinc sulphate — Oral syrup zinc sulphate
  Arms: Malnourished children
Other: Placebo — Oral syrup placebo
  Arms: Normal children

SUMMARY:
Zinc supplementation effect on appetite and growth of malnourished children

DETAILED DESCRIPTION:
The investigators will do s. Zinc and letting before and after zinc supplementation

ELIGIBILITY:
Inclusion Criteria:

* primary malnourished

Exclusion Criteria:

* zinc supplementation in the previous 3 months Children with chronic disease

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2017-09-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Appetite | From start of supplementation to the end of the three months of supplementation
  Child eating behavior questionnaire

SECONDARY OUTCOMES:
Weight | From start of supplementation to the end of the three months of supplementation
  Weight
Height | From start of supplementation to the end of the three months of supplementation
  Height

CONTACTS AND LOCATIONS:
Overall Officials: Marian Girgis, Principal Investigator — Ain Shams University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Imdad A, Rogner J, Sherwani RN, Sidhu J, Regan A, Haykal MR, Tsistinas O, Smith A, Chan XHS, Mayo-Wilson E, Bhutta ZA. Zinc supplementation for preventing mortality, morbidity, and growth failure in children aged 6 months to 12 years. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD009384. doi: 10.1002/14651858.CD009384.pub3. PMID 36994923